CLINICAL TRIAL: NCT04620083
Title: Effects of an Integrative Learning Program on Community Dwelling Old People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: Guangzhou Medical University (Other); Guangzhou University of Chinese Medicine (Other); Tung Wah College (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Hong Kong Nang Yan College of Higher Education (Other); Ginger Knowledge Transfer and Consultancy Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020_CTS001
Record Dates: First submitted 2020-10-29; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Dementia
Keywords: Dementia; Neuroplasticity; Integrative Learning; Slow Stream Rehabilitation; Novice-expert Continuum; Community Dwelling Old People
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: The research team randomly allocated the elderly to the control group (Con), Experimental 3-day normal group (Exp-N) and Experimental 5-day intensive group (Exp-I). For the control group, the participants received conventional therapy which included group activities for reality orientation, reminiscence therapy and activities organized by occupational therapists one hour a day, five days a week. In addition to conventional therapy, the two experimental groups also joined the integrative learning program. For consistency, Day 1 and 3 of the 3-day protocol were replicated as Day 4 and Day 5 of the 5-day protocol.
Who Masked: Investigator
Masking Description: Allocation concealment was done to avoid selection bias while blinding was done to research assistant who performed data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): For the control group, the participants received conventional therapy which included group activities for reality orientation, reminiscence therapy and activities organized by occupational therapists one hour a day, five days a week.
- Experimental 3-day Normal Group (Experimental): In addition to conventional therapy, the participants in this experimental groups also joined the integrative learning program for 3 days per week.
  Interventions: Other: Integrative Learning Program for Old People with Dementia
- Experimental 5-day Intensive Group (Experimental): In addition to conventional therapy, the participants in this experimental groups also joined the integrative learning program for 5 days per week. For consistency, Day 1 and 3 of the 3-day protocol were replicated as Day 4 and Day 5 of the 5-day protocol.
  Interventions: Other: Integrative Learning Program for Old People with Dementia

INTERVENTIONS:
Other: Integrative Learning Program for Old People with Dementia — The program included modalities for reality orientation, daily living skills training, reminiscence therapy, multisensory stimulation, fall prevention program, mindfulness activities, Meridian exercise, brain health program (Four Arts of the Chinese Scholar which referred to zither, go, calligraphy and painting) and health education. It was also agreed that case managers, caregivers, and participants were free to choose these treatments or could be assigned to a treatment regime on a 'mix and match' basis to suit their personality traits for improving their abilities to meet their own needs. This program was developed by the team using Delphi technique.
  Arms: Experimental 3-day Normal Group; Experimental 5-day Intensive Group

SUMMARY:
Objectives: To develop an integrative learning program and evaluate its effect on people with dementia. Methods: The study started from January 2017 to March 2018 and consisted of two stages. The first stage employed Delphi technique while the second an experimental design. An expert panel was invited to develop the integrative learning program based on the neuroplasticity and learning framework in the first stage. A mixed method approach was adopted for the evaluation of the program in the second stage. Questionnaires and clinical instruments were used to collect quantitative data. For qualitative data, verbatim transcripts of case conferences were coded, analyzed, and collapsed into themes and sub-themes by consensus. Results: Quantitatively, significant improvements in the participants' functional performance and well-being in the experimental groups, while qualitatively, improvements on their communications, emotions, connectedness with self and others, and well-being. Conclusion: Overall the evaluation was positive; however, larger sample size of old people from more community care centers would provide more conclusive results.

DETAILED DESCRIPTION:
Stage 1 - The development of the integrative learning program

Delphi technique was employed to gain consensus in the best possible therapeutic interventions for old people with dementia among members of the expert panel. The panel consisted of 8 health professionals including a gerontic care nurse, a registered nurse, an occupational therapist, a physiotherapist, a Chinese medicine practitioner, a mindfulness practitioner, a nutritionist, and a neuroscientist. They all had more than 10 years of experience in their own disciplines.

A research team member explained to the experts individually the purpose of having the Panel and the importance of opinion sharing and idea exchange. Subsequent exchanges covered the conceptual framework, needs of people with dementia, components of the program operation and the intervention protocol. The experts did not meet but to provide their views through emails or audio recordings. Research members organized, collated the views, presented the aggregated views iteratively to each expert for consideration. The exchange on each topic terminated when all experts reached total agreement on their analysis and views were exhausted. Upon completion of each round, a summary was sent to all experts for accuracy checking. With this iterative approach, 12 rounds of exchange were necessitated to develop the complete integrative learning protocol.

To dispel any unrealistic expectations and facilitate learning, training in goal setting skills is needed in the integrative learning program. It was agreed among the experts that people with dementia have different needs and expectations, and various levels of difficulty and ability to meet them, be it basic (novice) or advanced (expert). Hence the Panel formulated a list of developmental needs which are necessary and essential for quality living of people with dementia. The goal of development of each need was also identified based on a novice-expert continuum and the conceptual framework of neuroplasticity and learning.

The Panel reviewed some common dementia management programs used in local institutions. Although these programs have included many contemporary treatment modalities, the results were not marked. The Panel also commented that the treatment modalities could have been sufficient but the piece-meal approach might undermine their efficacy. They concluded that an integrated and structured multi-modality approach together with emotion management should be adopted for the integrative learning program. The multi-modality treatments in the program were structured sessions that employed physical, cognitive, social, and emotional stimulations to intervene dementia. The modalities selected for the program included reality orientation, daily living skills training, reminiscence therapy, multisensory stimulation, fall prevention program, mindfulness activities, Meridian exercise, brain health program (Four Arts of the Chinese Scholar which referred to zither, go, calligraphy and painting) and health education. It was also agreed that case managers, caregivers, and participants were free to choose these treatments or could be assigned to a treatment regime on a 'mix and match' basis to suit their personality traits for improving their abilities to meet their own needs.

Based on the outcome of the above Delphi exercise, the experts brain-stormed the contents and details of each, followed by discussions before resolutions were made by consensus. Consensus was reached for the duration of a standard 3-day protocol and 5-day protocol. The 5-day protocol was an extended version of the 3-day one which allowed the participants to practice more in a designated time. Table 2 shows the 3-day integrative learning protocol. Interventions using the protocol were carried out by case managers who could be nurses, occupational therapists, or other health professionals. These case managers were independent of the research team. To ensure the competency of the case managers, each one had to attend a 3-day training workshop, with one day on theories, another day on practical training by 3 members of the Expert Panel (the gerontic care nurse, the nurse, and the occupational therapist) and the final day on quality assurance.

Stage 2 - Proof of concept: The evaluation of the implementation of the developed program by using a mixed method approach

i) Quantitative Method The study was held in three community care centers run by the same non-profit organization (NPO) and their routine and care provided were the same across their centers. Two types of services were provided in community care centers, residential and day care. The centers were located in different districts where residents were in public housing. Three centers were randomly drawn from the NPO by drawing lots. Eligible older people with dementia from the centers were recruited by convenience sampling. All participants continued with their daily routines and medications during the research period.

Having received consent from both the eligible older people and their relatives, the research team randomly allocated them to the control group (Con), Experimental 3-day normal group (Exp-N) and Experimental 5-day intensive group (Exp-I). For the control group, the participants received conventional therapy which included group activities for reality orientation, reminiscence therapy and activities organized by occupational therapists one hour a day, five days a week. In addition to conventional therapy, the two experimental groups also joined the integrative learning program. For consistency, Day 1 and 3 of the 3-day protocol were replicated as Day 4 and Day 5 of the 5-day protocol.

Allocation concealment was done to avoid selection bias while blinding was done to research assistant who performed data collection. Data were collected before the start of the program (T0) and upon its completion (T2 - at 6th month) for all 3 groups. For the two experimental groups, there was a mid-intervention evaluation (T1- at 3rd month). During the intervention, the trained case managers evaluated the conditions of the participants on a monthly basis until the completion of the program. They joined the monthly case conferences held by the respective centers listening to progress of the participants reported by center staff.

With the adoption of the mixed method approach, quantitative data were collected using 10 validated clinical test instruments while qualitative data were based on the verbatim transcripts of the monthly case conferences.

ii) Qualitative Method For the qualitative data, the verbatim transcripts of the case conferences were used for thematic analysis. These verbatim records were transcribed and coded for content analysis, based on the conceptual framework of the integrative learning program. The research assistant first identified words /segments in each transcript and then condensed them into meaningful units. Two panel members abstracted all the condensed meaning units into subthemes.

ELIGIBILITY:
Inclusion Criteria:

* People aged 65 or above
* Members of the community care centers
* Diagnosed with dementia and mild cognition impairment (determined by the Montreal Cognitive Assessment Test for Dementia, MoCA score 12.7-20.1 depending on education level)

Exclusion Criteria:

* Living alone
* With communication difficulties like language barriers, deafness, dysphasia and/or severe dysarthria
* Recently participated in another dementia program
* With known history of psychotic illnesses such as schizophrenic, psychiatric, or with organic brain diseases such as brain tumors

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline disability level due to dementia at 3 months | Up to 3 months
  By Functional Assessment Stage Test, the minimum is Stage 1 (Normal Aging) and the maximum is Stage 7f (Severe Dementia), the lower is the better
Change from baseline disability level due to dementia at 6 months | Up to 6 months
  By Functional Assessment Stage Test, the minimum is Stage 1 (Normal Aging) and the maximum is Stage 7f (Severe Dementia), the lower is the better
Change from baseline cognitive function impairment due to dementia at 3 months | Up to 3 months
  By Montreal Cognitive Assessment - Hong Kong Version, the minimum is 0 score and the maximum is 30, a score of 26 or over is considered to be normal, the higher is the better
Change from baseline cognitive function impairment due to dementia at 6 months | Up to 6 months
  By Montreal Cognitive Assessment - Hong Kong Version, the minimum is 0 score and the maximum is 30, a score of 26 or over is considered to be normal, the higher is the better

SECONDARY OUTCOMES:
Change from baseline functional independence at 3 months | Up to 3 months
  By Barthel Index, the minimum is 0 score and the maximum is 20, the higher is the better
Change from baseline functional independence at 6 months | Up to 6 months
  By Barthel Index, the minimum is 0 score and the maximum is 20, the higher is the better
Change from baseline mobility function at 3 months | Up to 3 months
  By Timed Up and Go Test, below 12 seconds is considered to be normal performance, the shorter is the better
Change from baseline mobility function at 6 months | Up to 6 months
  By Timed Up and Go Test, below 12 seconds is considered to be normal performance, the shorter is the better
Change from baseline static balance and fall risk at 3 months | Up to 3 months
  By Berg Balance Test, the minimum is 0 score and the maximum is 56, the higher is the better
Change from baseline static balance and fall risk at 6 months | Up to 6 months
  By Berg Balance Test, the minimum is 0 score and the maximum is 56, the higher is the better
Change from baseline abnormal cognitive function in elderly at 3 months | Up to 3 months
  By Abbreviated Mental Test, the minimum is 0 score and the maximum is 10, the higher is the better
Change from baseline abnormal cognitive function in elderly at 6 months | Up to 6 months
  By Abbreviated Mental Test, the minimum is 0 score and the maximum is 10, the higher is the better
Change from baseline depression in elderly at 3 months | Up to 3 months
  By Geriatric Depression Scale, the minimum is 0 score and the maximum is 30, the lower is the better
Change from baseline depression in elderly at 6 months | Up to 6 months
  By Geriatric Depression Scale, the minimum is 0 score and the maximum is 30, the lower is the better
Change from baseline quality of life in Alzheimer's Disease at 3 months | Up to 3 months
  By the scale Quality of Life - Alzheimer's Disease, the minimum is 0 score and the maximum is 52, the higher is the better
Change from baseline quality of life in Alzheimer's Disease at 6 months | Up to 6 months
  By the scale Quality of Life - Alzheimer's Disease, the minimum is 0 score and the maximum is 52, the higher is the better
Change from baseline communication abilities at 3 months | Up to 3 months
  By Holden Communication Scale, the minimum is 0 score and the maximum is 48, the lower is the better
Change from baseline communication abilities at 6 months | Up to 6 months
  By Holden Communication Scale, the minimum is 0 score and the maximum is 48, the lower is the better
Change from baseline mental well-being at 3 months | Up to 3 months
  By World Health Organization (Five) Well-Being Index, the minimum is 0 score and the maximum is 25, the higher is the better
Change from baseline mental well-being at 6 months | Up to 6 months
  By World Health Organization (Five) Well-Being Index, the minimum is 0 score and the maximum is 25, the higher is the better

CONTACTS AND LOCATIONS:
Locations (1):
- The Education University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No